CLINICAL TRIAL: NCT00686036
Title: A Randomized, Double-blind, Multicentre, Phase II Controlled Trial Assessing ZACTIMATM (Vandetanib) Against Placebo in Prolonging the Off-treatment Interval in Prostate Cancer Subjects Undergoing Intermittent Androgen Deprivation Hormonal Therapy
Brief Title: Trial Assessing Zactima Against Placebo in Prostate Cancer Subjects Undergoing Intermittent Androgen Deprivation Hormonal Therapy
Acronym: ZENITH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4200L00010
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Results first posted 2011-05-24 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; hormone treatment
MeSH Terms: conditions — Prostatic Neoplasms | interventions — vandetanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vandetanib (Experimental): 300 mg orally, once daily for up to 18 months
  Interventions: Drug: vandetanib
- Placebo (Placebo Comparator): orally, once daily for up to 18 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: vandetanib — 300 mg orally, once daily for up to 18 months
  Other Names: Zactima
  Arms: vandetanib
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether treatment with Zactima for up to 18 months will prolong the off-treatment interval in patients who are undergoing intermittent androgen deprivation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate cancer
* Prostate specific antigen (PSA) greater than or equal to 5 ng/mL
* Recent completion of first hormone treatment [intermittent androgen deprivation with a Luteinising hormone releasing hormone (LHRH) analogue]
* Screening PSA ≤1.0 ng/mL (within 6 weeks prior to study Day1)

Exclusion Criteria:

* Bone or soft tissue metastases
* Significant cardiovascular disease including hypertension not controlled by medical therapy or history of irregular heart beats or recent heart attack

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-05; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (11):
- Canada (11):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Victoria, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Granby

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 25 male patients signed informed consent at 12 centres in Canada between May 2008 and February 2010. Out of these 25 patients, 17 patients were randomized with 9 patients in the vandetanib treatment arm and 8 patients in the placebo arm.
Pre-assignment Details: To be eligible for enrollment into the study, patients had to have received treatment with ADT for 36 weeks (± 4 weeks), with a pre-ADT PSA ≥ 5 ng/mL. Also, they should have had a screening PSA ≤ 1.0 ng/mL (within 6 weeks prior to study Day 1)
Groups:
- Vandetanib: Vandetanib 300 mg tablet
- Placebo: Placebo to match vandetanib 300 mg tablet
Period: Overall Study
Arm/Group | Vandetanib | Placebo
Started | 9 | 8
Completed | 0 | 2
Not Completed | 9 | 6
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Study terminated by AstraZeneca | 2 | 1
Not completed — PSA ≥ 10ng/mL | 1 | 0
Not completed — Other reasons not identified | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vandetanib | Placebo | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72 (7.263) | 71.5 (7.709) | 71.5 (7.489)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 9 | 8 | 17
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Not Reaching a PSA ≥ 5ng/mL by 52 Weeks During the Off-treatment Phase of Androgen Deprivation Therapy (ADT)
Time Frame: 52 weeks
Population: Due to slow recruitment, the study was terminated early. Efficacy analysis was not performed. Therefore, zero participants were analyzed.
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants Not Reaching PSA ≥ 5ng/mL and/or PSA 10ng/mL (Biochemical Failure) by 78 Weeks During the Off-treatment Phase of Androgen Deprivation Therapy (ADT)
Time Frame: 78 weeks during off-treatment phase of ADT
Population: as for outcome 1
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to PSA Progression (PSA ≥ 5ng/mL and PSA ≥ 10ng/mL)
Time Frame: From the time o PSA rise from the date of randomization to both PSA ≥ 5ng/mL and PSA ≥ 10ng/mL
Population: as for outcome 1
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Serum Testosterone Levels
Time Frame: Change from baseline at each visit post-randomization until until week 78
Population: as for outcome 1
Arm/Group | Vandetanib | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Vandetanib | Placebo
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/8
Other Adverse Events (participants affected / at risk) | 9/9 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib (N=9) | Placebo (N=8)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis Viral (Infections and infestations) | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
Alanine aminotrasferase increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib (N=9) | Placebo (N=8)
Diarrhoea (Gastrointestinal disorders) | 7 | 2
Nausea (Gastrointestinal disorders) | 3 | 2
Fatigue (General disorders) | 2 | 3
Oedema peripheral (Gastrointestinal disorders) | 2 | 3
Nasopharyngitis (Infections and infestations) | 2 | 3
Electrocardiogram QT prolonged (Investigations) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Dizziness (Nervous system disorders) | 3 | 1
Listless (Psychiatric disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0
Chills (General disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 2 | 0
Hot flush (Vascular disorders) | 1 | 2
Pallor (Vascular disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 1
Hepatic Lesion (Hepatobiliary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Carbuncle (Infections and infestations) | 0 | 1
Helicobacter infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 0 | 1
Tinea cruris (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Cardiac Murmur (Investigations) | 0 | 2
Weight decreased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Amnesia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0
Renal Cyst (Renal and urinary disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0

LIMITATIONS AND CAVEATS:
It was planned that approx 100 patients would be recruited over a period of approx 2 years, due to slow recruitment the study was terminated early. No statistical analyses was done and no conclusion can be drawn about the outcomes in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.